CLINICAL TRIAL: NCT02623621
Title: A Single-arm Phase II Study of Circulating Soluble Vascular Endothelial Growth Factor Receptor 2 (VEGFR-2) as Predictor of Benefit From Bevacizumab (Bev) Beyond Progression in Metastatic Colorectal Cancer (mCRC) - the CIRCUS Study
Brief Title: Soluble Vascular Endothelial Growth Factor Receptor 2 as Predictor of Benefit From Bevacizumab Beyond Progression in Metastatic Colorectal Cancer
Acronym: CIRCUS
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Alfredo Falcone, MD, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: CIRCUS
Record Dates: First submitted 2015-12-01; First posted 2015-12-08 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Paired plasma and blood samples will be collected at baseline, at the time of every disease assessment and at the time of disease progression
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: chemotherapy plus bevacizumab — Every chemotherapy regimen combined with bevacizumab is allowed

SUMMARY:
A growing amount of reports has consistently evidenced that a sustained inhibition of the angiogenesis is an effective therapeutic strategy, able to improve the outcome of metastatic colorectal cancer (mCRC) patients.

In the last decade different biologic agents targeting angiogenesis have been approved for the treatment of mCRC, such as bevacizumab, aflibercept and regorafenib, and, more recently, solid evidences have demonstrated the efficacy of a sustained antiangiogenic approach even beyond the first progression to a bevacizumab-containing regimen. In particular, two phase III randomized trials proved the effectiveness of prosecuting bevacizumab in second-line switching the chemotherapeutic regimen in patients already treated with bevacizumab in first-line. Preliminary experiences evidenced that circulating levels of angiogenesis-related markers are significantly modulated during first-line chemotherapy plus bevacizumab. In particular, a wide variability of plasma soluble Vascular Endothelial Growth Factor Receptor-2 (VEGFR-2) levels is observed at the time of disease progression and retrospective data suggest that benefit from the continuation of bevacizumab may be restricted to patients with high levels of soluble VEGFR-2 at the first evidence of disease progression. This study aims at prospectively validating those retrospective data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of ≥ 18 years of age
* Progressive disease during or after first-line chemotherapy plus bevacizumab, including fluoropyrimidine alone (5-fluorouracil or capecitabine), fluoropyrimidine in combination with oxaliplatin (XELOX or FOLFOX regimen) or irinotecan (FOLFIRI regimen) or with oxaliplatin and irinotecan (FOLFOXIRI regimen);
* No more than 3 months from the last administration of bevacizumab and evidence of progressive disease are allowed;
* Measurable disease according to RECIST 1.1.
* Indication to second-line treatment with a bevacizumab-containing second-line regimen (second-line XELOX, FOLFOX, FOLFIRI and FOLFOXIRI plus bevacizumab are allowed);
* Neutrophils 1.5 x 109/L, Platelets 100 x 109/L, Hgb >9 g/dl
* Total bilirubin 1.5 time the upper-normal limits (UNL) of the institutional normal values and ASAT (SGOT) and/or ALAT (SGPT) 2.5 x UNL, or 5 x UNL in case of liver metastases, alkaline phosphatase 2.5 x UNL, 5 x UNL in case of liver metastases
* Creatinine clearance >50 mL/min or serum creatinine 1.5 x UNL
* Urine dipstick of proteinuria <2+. Patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate <1 g of protein/24 hr
* Will and ability to comply with the protocol
* Written informed consent to study procedures.

Exclusion Criteria:

* Patient unable to give consent
* Absolute contraindications to the use of bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mCRC progressed on or after a 1st-line bevacizumab-containing regimen and candidate to continue bevacizumab beyond progression, in combination with a 2nd-line chemotherapy regimen.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2015-11; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | from treatment start until disease progression, according to RECIST 1.1, or death due to any cause, whichever occurs first, up to 12 months after last patient last visit

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, PI, Italy